CLINICAL TRIAL: NCT00508612
Title: Impact of LifeSkills Training on Blood Pressure in Youth
Brief Title: Effectiveness of an Anger and Stress Management Program on Reducing Blood Pressure Levels in Youth
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Collaborators: Williams LifeSkills (Industry)
Responsible Party: Principal Investigator, Assistant Professor, National Heart, Lung, and Blood Institute (NHLBI)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 497; R42HL072644-02A2 (NIH)
Record Dates: First submitted 2007-07-27; First posted 2007-07-30 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2013-03

CONDITIONS: Cardiovascular Diseases; Hypertension
Keywords: Blood Pressure; Systolic Blood Pressure; Diastolic Blood Pressure; Ambulatory Blood Pressure Monitoring; Relaxation; Meditation; Coping Skills; Adolescents
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): The 12-lesson Williams LifeSkills anger and stress management workshop (WLS) enhances awareness of thoughts and feelings in stressful situations, and provides training in evaluation, deflection, problem-solving, assertion, saying no, speaking, listening, empathy, and emphasizing positives.
  Interventions: Behavioral: Williams LifeSkills Stress and Anger Management Workshop
- 2 (Placebo Comparator): Control group (will attend regular high school classes)
  Interventions: Behavioral: High school classes

INTERVENTIONS:
Behavioral: Williams LifeSkills Stress and Anger Management Workshop — Williams LifeSkills Stress and Anger Management Workshop
  Arms: 1
Behavioral: High school classes — The control group will attend regular high school classes.
  Arms: 2

SUMMARY:
High blood pressure can often be caused by stress or anxiety. This study will evaluate a school-based stress and anger management program that aims to lower blood pressure and anger levels among high school students.

DETAILED DESCRIPTION:
High blood pressure can be caused by many factors, including stress, anxiety, diabetes, kidney disease, or obesity. In many people, there is no identifiable cause for their high blood pressure; this is known as essential hypertension (EH). Increasingly, children are being diagnosed with high blood pressure, which may lead to an increased risk of developing EH as adults. Therefore, the need exists for an effective blood pressure reduction program targeted toward youth. Research has shown that improving people's abilities to manage stress and anger reduces their risk of developing high blood pressure and heart disease. The Williams LifeSkills (WLS) workshop is a program that teaches people to cope with stressful situations. It has been shown to improve heart health, including blood pressure levels, in adults with cardiovascular disease. However, the effect of stress and anger management programs on blood pressure levels in youth has not been widely studied. Study researchers have developed and preliminarily tested a school-based anger and stress management WLS program. This study will evaluate the effectiveness of the school-based WLS program at reducing blood pressure and anger levels in high school students. If successful, this program could be implemented in schools across the country.

This study will enroll high school students. Participants will be randomly assigned to either a 12 lesson WLS program or a control group. Participants in the control group will attend regular high school classes. Participants in the WLS program will attend 12 sessions that will focus on coping skills to help manage stress and anger levels. At baseline, the end of the 12 lesson program, and follow-up visits 3 and 6 months later, participants will complete questionnaires on anger levels; life skills; hostility; stress; self-esteem; and attitudes toward school, teachers, and parents. They will also wear a blood pressure monitor for a 24-hour period.

ELIGIBILITY:
Inclusion Criteria:

* High school student

Exclusion Criteria:

* History of any chronic illness or any chronic health problem requiring pharmacological treatment (e.g., asthma, sickle cell disease, epilepsy)
* Adolescents with ambulatory systolic blood pressure greater than the 95th percentile based on age, sex, and height at screening will be allowed to participate in the workshop but may be excluded from testing
* Unwilling to be assigned into a specific treatment group

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 259 (Actual)
Dates: Start 2007-04; Primary Completion 2009-05 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Reduction in day-time ambulatory systolic blood pressure | Measured at post-intervention after the 12 lesson program and at 3- and 6-month follow-up visits

CONTACTS AND LOCATIONS:
Overall Officials: Vernon A. Barnes, PhD, Principal Investigator — Medical College of Georgia - Georgia Prevention Institute; Virginia P. Williams, PhD, Principal Investigator — Williams LifeSkills
Locations (3):
- United States (3):
  - Richmond County Board of Education Public Schools, Augusta, Georgia
  - Medical College of Georgia - Georgia Prevention Institute, Augusta, Georgia
  - Williams LifeSkills, Durham, North Carolina

REFERENCES:
- [Result] Barnes VA, Williams VP, Williams RB. Impact of Williams LifeSkills training on blood pressure in adolescents. Psychosomatic Medicine. 2005;67:A78.
- [Result] Barnes VA, Williams VP, Williams RB. Effects of Williams LifeSkills training on anger reduction in African American adolescents. Psychosomatic Medicine. 2005;67:A53.
- [Result] Barnes VA, Williams VP, Williams RB, Johnson MH, Stevens AM, Shenbagarajan VP. Effect of Williams Lifeskills training on anger control in African American adolescents (abstract 014). Paper presented at: ISHIB2008: 23rd Annual International Interdisciplinary Conference on Hypertension and Related Cardiovascular Risk Factors in Ethnic Populations, 2008; New Orleans, LA.
- [Result] Barnes VA, Williams VP, Williams RB, Johnson MH, Murrell AS, Shenbagarajan VP, Dubert C. Williams Lifeskills® training lowers school-time ambulatory blood pressure in adolescents. Paper accepted for presentation at: Society of Behavioral Medicine Annual Meeting April 22-25, 2009; Montreal, Canada.
- [Result] Barnes VA, Williams VP, Williams RB, Shenbagarajan VP, Bentley DR, Johnson MH. Effect of Williams Lifeskills Training on Anger and Anxiety in Adolescents. Psychosomatic Medicine. 2010;72(3):A70.
- See also: website about Williams LifeSkills — http://www.williamslifeskills.com/